CLINICAL TRIAL: NCT00484783
Title: Prospective Evaluation of the Intraoperative Use of Translumenal Flexible Endoscopes During Combined Flexible and Laparoscopic Foregut and Urologic Surgery
Brief Title: Transluminal Flexible Endoscopic Procedure in Foregut and Urologic Surgery
Acronym: NOTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, Prinicpal Investigator, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-06-13
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Gastric Foreign Body, Nos; Disorder of Abdomen (Disorder); Foreign Body in Esophagus; Prostatic Diseases; Disease of Small Intestine
Keywords: Laparoscopic Surgical Procedures; Endoscopic Surgical Procedures; Laparoscopic & endoscopic procedures with a gastrotomy; or opening in bladder or urethra
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Prostatic Diseases | interventions — Natural Orifice Endoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prospective (Experimental): Subjects scheduled to receive procedure
  Interventions: Procedure: Natural Orifice Transluminal Endoscopic Surgery (NOTES)
- Historical (Other): Chart review control group
  Interventions: Procedure: Natural Orifice Translumenal Endoscopic Surgery (NOTES)

INTERVENTIONS:
Procedure: Natural Orifice Transluminal Endoscopic Surgery (NOTES) — Patients will have the standard laparoscopic procedure and the NOTES procedure will be added. The surgical procedure will require two operating teams: one led by a laparoscopic surgeon, the other by an endoscopic surgeon. During the usual course of the surgery, the flexible endoscope will be passed through the mouth urethra top gain access to the peritoneal cavity.
  Other Names: NOTES Surgery
  Arms: Prospective
Procedure: Natural Orifice Translumenal Endoscopic Surgery (NOTES) — chart review of historical data from control group
  Other Names: NOTES Surgery
  Arms: Historical

SUMMARY:
NOTES access is safe and feasible in the controlled human setting and comparable to standard-of-care surgical techniques. NOTES exploration of the abdomen provides adequate visualization comparable to laparoscopy.

DETAILED DESCRIPTION:
This is a prospective clinical trial to evaluate the feasibility of obtaining peritoneal cavity access from natural orifice translumenal endoscopic surgery (NOTES) during combined laparoscopic-endoscopic foregut surgery. Post-operative course will be compared with a historical chart-review control group of patients undergoing standard laparoscopic foregut and urologic surgery.

The study group will be compiled by open enrollment for male and female adult subjects scheduled for combined laparoscopic-endoscopic surgery of the stomach, abdominal esophagus, prostate, bladder, proximal small intestine or who meet inclusion and exclusion criteria. The historical chart-review control group will be randomly chosen from patients from 2003-2006 having undergone combined laparoscopic-endoscopic surgery of the foregut, prostate, or bladder and as determined by CPT coding.

The purpose of the study is to determine if NOTES access and abdominal exploration is feasible, safe, offers comparable visualization to laparoscopy in a controlled human setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an already combined laparoscopic and endoscopic foregut procedure with general anesthesia
* Patients undergoing a prostatectomy or cystectomy with general anesthesia
* All patients will have a planned gastrotomy for exploration, foreign body removal, or removal of tissue, making it a contaminated case or a planned cystotomy or urethrotomy for exploration, foreign body removal or removal of tissue such as prostatectomy or bladder resection.
* No overwhelming medical co-morbidities
* Subject is 18 years of age or older
* Subject is his or her own medical decision maker
* Subject agrees to participate, fully understands content of informed consent form, and signs the informed consent form

Exclusion Criteria:

* Patients undergoing a non-palliative procedure in the face of resectable adenocarcinoma of the foregut or genitourinary tract
* Linitis Plastica
* Evidence of Active Bowel Obstruction
* Patients with history of oropharyngeal, esophageal, or gastric adenocarcinoma.
* Esophageal stricture prohibiting passage of an endoscope
* Urethral stricture prohibiting passage of an endoscope
* Emergent Surgery
* At any time during pre-operative or intra-operative periods, evidence of unresectability is demonstrated
* Any intra-operative condition prior to surgical resection that results in abortion of the surgical procedure
* Any contraindication to surgery
* Pregnancy or actively breastfeeding women
* Prisoners or Wards of State

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
30 day Post-op NOTES feasibility outcomes: | 30 days post-op
  * Number of successful NOTES access attempts
  * Number of failed NOTES access attempts
  * Injury to collateral organs or structures
  * Time to gain access to peritoneal cavity
  * Necessary balloon dilator size required for translumenal passage of endoscope

SECONDARY OUTCOMES:
30 Day Post-OP Evaluation of Efficacy of NOTES access when compared to historical control groups undergoing laparoscopic access during foregut surgery | 30 Day Post-OP
  Description: Mortality Post-Op Mobidity repeat sugery Intra-Op or Post-Op RBC Transfusion Intra-Abdominal Abscess Superficial Surgical Site Infection Antibiotics>24th Post-Op
  Safety Issue?: Yes
30 Day NOTES Post - Op Evaluation of Adequacy of Abdominal Exploration | 30 Day Post - Op
  Description: Identification of Specified Abdominal and Pelvic Organs Time to Adequately Visualize Specified Abdominal and Pelvic Organs Comparitive findings between standardaized abdominal exploration between laparoscopy and NOTES techniques

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Marks, MD, Principal Investigator — University Hospitals of Cleveland/ Institute for Surgical Innovation
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States